CLINICAL TRIAL: NCT05568147
Title: A Prospective Multicenter Clinical Study of Aspirin for Prophylaxis in Patients With Hereditary or Acquired Thrombotic Thrombocytopenic Purpura
Brief Title: Aspirin for Prophylaxis of TTP
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, HAN Yue, vice director hematologic department, The First Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SOOCHOW-HY-2022-11
Record Dates: First submitted 2022-09-25; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Thrombotic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aspirin 100 mg daily (Experimental): Once enrolled, patients will receive aspirin 100mg orally once per day
  Interventions: Drug: Aspirin tablet
- Placebo (Placebo Comparator): Once enrolled, patients will receive placebo orally once per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin tablet — When patients are randomized into the intervention group, they will receive aspirin at the dosage of 100mg orally once every day.
  Arms: Aspirin 100 mg daily
Drug: Placebo — When patients are randomized into the placebo group, they will receive placebo orally once a day.
  Arms: Placebo

SUMMARY:
Thrombotic thrombocytopenic purpura (TTP) is a rare and life-threatening thrombotic microangiopathy characterized by thrombocytopenia, microangiopathic hemolytic anemia, and microvascular thrombosis causing neurological and renal abnormalities; it is associated with massive depletion of platelets in the microvasculature to form microthrombi1 . Long-term follow-up of patients with congenital TTP (cTTP) revealed frequent strokes and renal injury. Of 217 surviving patients, 62 (29%) had a stroke; the median age was 21 years. iTTP patients also require long-term follow-up. iTTP patients with low ADAMTS13 activity (<70%) in remission have a 28% risk of stroke. Survival rates of iTTP patients in remission were lower than those of age-, race-, and sex-matched populations. In terms of stable treatment, maintenance therapy is not recommended for patients with iTTP. Previous studies have shown that aspirin may be able to prevent stroke complications in patients with cTTP and iTTP. In addition to its potential efficacy, the risks of aspirin are small and inexpensive. Aspirin is very effective in secondary prevention of stroke 6. However, the therapeutic value of aspirin in TTP has not been studied previously. To improve the prognosis and survival of patients with cTTP and iTTP, we propose to conduct a prospective study to observe the efficacy and safety of aspirin in patients with cTTP and iTTP in remission.

DETAILED DESCRIPTION:
Thrombotic thrombocytopenic purpura (TTP) is a rare, life-threatening thrombotic microangiopathy. It is characterized by thrombocytopenia, microangiopathic hemolytic anemia, and microvascular thrombosis causing neurologic and kidney abnormalities . TTP is caused by a severe deficiency of ADAMTS13 (A Disintegrin and Metalloprotease with ThromboSpondin type 1 repeats, member 13) . Severe ADAMTS13 deficiency can be hereditary (hTTP), caused by biallelic pathogenic mutations of the ADAMTS13 genes, or acquired (iTTP), caused by anti-ADAMTS13 autoantibodies. Its main diagnostic criterion is a severe deficiency of ADAMTS13 (activity <10%) .

hTTP is currently managed by prophylaxis with plasma infusions. Because lifetime plasma infusions are a major lifestyle burden, the current practice is to begin prophylaxis when ischemic symptoms occur. Evaluation of plasma prophylaxis by the International Hereditary Registry reported that it was not effective for decreasing the occurrence of acute episodes. When recombinant ADAMTS13 (rADAMTS13) is commercially available, prophylaxis may begin sooner and be more effective. Acute episodes of iTTP are effectively treated with ADAMTS13 replacement and immunosuppression. During remission, immunosuppression is recommended to prevent relapse if ADAMTS13 activity is <20%. If ADAMTS13 activity is less than normal but ≥20%, no treatment is recommended.

Long-term follow-up of patients with hTTP has identified the frequent occurrence of stroke and kidney injury. Among 217 patients who survived infancy, 62 (29%) had had a stroke; the median age was 21 years. Long-term follow-up is also required for patients with iTTP. iTTP patients with low ADAMTS13 activity (<70%) during remission have a 28% risk for stroke. Survival of iTTP patients in remission is less than the age, race, and gender-match population. No maintenance treatment is recommended for patients with iTTP.

Severe ADAMTS13 deficiency in patients with TTP allows the circulation of ultra-large multimers of von Willebrand factor (VWF). Turbulent circulation causes exposure of the VWF platelet binding site. Binding of the platelet VWF receptor, GPIbα, to the ultra-large VWF multimers is the essential initial which step for the initiation of thrombosis. A recent study documented that platelet binding to von Willebrand factor activates the platelet fibrinogen receptor, αIIbβ3, initiating platelet aggregation. Aspirin blocks αIIbβ3 activation and prevents platelet aggregation. Studies of TTP in mice have documented that aspirin decreases thrombosis. These data suggest that it may provide protection against stroke in patients with hTTP and iTTP. In addition to its potential efficacy, aspirin has minimal risks, and it is inexpensive.

Aspirin is very effective for the secondary prevention of stroke. However, the therapeutic value of aspirin in TTP has not previously been studied.

To improve the prognosis and survival of patients with hTTP and iTTP, we propose to conduct a prospective study to observe the efficacy and safety of aspirin in patients with the iTTP and hTTP in remission.

ELIGIBILITY:
Inclusion Criteria:

1. Those who voluntarily signed the informed consent form and were able to comply with the study protocol.
2. Subjects diagnosed with severe ADAMTS13 deficiency, defined as ADAMTS13 activity <10%, documented in the patient's medical history or at screening. Note: In patients receiving fresh frozen plasma (FFP) or other prophylactic treatments containing ADAMTS13 products, plasma ADAMTS13 activity levels at screening may exceed 10%. hTTP will be documented by ADAMTS13 activity <10% and biallelic pathogenic ADAMTS13 mutations. Patients with hTTP may be asymptomatic. iTTP will be diagnosed by ADAMTS13 activity <10% and the presence of an ADAMTS13 activity inhibitor (or comparable test for anti-ADAMTS13 antibodies). The diagnosis of hTTP may be supported by the recovery of ADAMTS13 activity to >10% during clinical remission.
3. Subjects do not exhibit any severe symptoms of TTP at the time of screening. At screening, patients with mild but stable laboratory abnormalities (LDH not higher than three times the upper limit of normal; platelet count not less than 100,000/microliter) are eligible for enrollment.
4. No stroke was detected on cranial MRI and there was no previous history of stroke.
5. The subject is willing and able to comply with the requirements of this protocol.

Exclusion Criteria:

1. Subject has a history of significant neurological events, such as a major stroke, indicating that a relapse may have serious consequences, as judged by the investigator
2. Subject has increased risk for bleeding (e.g., platelet count <30,000/µL, severe coagulopathy, gastrointestinal disease)
3. Subject has a history of drug and/or alcohol abuse within six months before enrollment.
4. Subject has a life expectancy of fewer than three months.
5. The investigator considers the subject unable or unwilling to cooperate with the study procedures.
6. The subject is a family member or employee of the investigator.
7. The patient is pregnant or breast-feeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with ischemic stroke | From first administration of aspirin to 3 years after treatment.
  Ischemic stroke was assessed with MRI imaging.

SECONDARY OUTCOMES:
Number of participants with relapse | From first administration of aspirin to 3 years after treatment.
  Relapse refers to the presence of TTP symptoms with less than 10% ADAMTS13 activity.
Number of participants with major bleeding | From first administration of aspirin to 3 years after treatment.
  Major bleedings refer to the heavy bleedings of the mains organs of the body, usually include intracranial bleeding and gastrointestinal bleeding et al.. Brain computed tomography and gastrointestinal endoscope are the common approaches for diagnosing major bleedings.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joly BS, Coppo P, Veyradier A. Thrombotic thrombocytopenic purpura. Blood. 2017 May 25;129(21):2836-2846. doi: 10.1182/blood-2016-10-709857. Epub 2017 Apr 17. PMID 28416507
- [Background] Levy GG, Nichols WC, Lian EC, Foroud T, McClintick JN, McGee BM, Yang AY, Siemieniak DR, Stark KR, Gruppo R, Sarode R, Shurin SB, Chandrasekaran V, Stabler SP, Sabio H, Bouhassira EE, Upshaw JD Jr, Ginsburg D, Tsai HM. Mutations in a member of the ADAMTS gene family cause thrombotic thrombocytopenic purpura. Nature. 2001 Oct 4;413(6855):488-94. doi: 10.1038/35097008. PMID 11586351
- [Background] Scully M, Yarranton H, Liesner R, Cavenagh J, Hunt B, Benjamin S, Bevan D, Mackie I, Machin S. Regional UK TTP registry: correlation with laboratory ADAMTS 13 analysis and clinical features. Br J Haematol. 2008 Sep;142(5):819-26. doi: 10.1111/j.1365-2141.2008.07276.x. Epub 2008 Jul 8. PMID 18637802
- [Background] Tsai HM. Thrombotic Thrombocytopenic Purpura: Beyond Empiricism and Plasma Exchange. Am J Med. 2019 Sep;132(9):1032-1037. doi: 10.1016/j.amjmed.2019.03.009. Epub 2019 Mar 28. PMID 30928346
- [Background] Shao B, Hoover C, Shi H, Kondo Y, Lee RH, Chen J, Shan X, Song J, McDaniel JM, Zhou M, McGee S, Vanhoorelbeke K, Bergmeier W, Lopez JA, George JN, Xia L. Deletion of platelet CLEC-2 decreases GPIbalpha-mediated integrin alphaIIbbeta3 activation and decreases thrombosis in TTP. Blood. 2022 Apr 21;139(16):2523-2533. doi: 10.1182/blood.2021012896. PMID 35157766
- [Background] Rothwell PM, Algra A, Chen Z, Diener HC, Norrving B, Mehta Z. Effects of aspirin on risk and severity of early recurrent stroke after transient ischaemic attack and ischaemic stroke: time-course analysis of randomised trials. Lancet. 2016 Jul 23;388(10042):365-375. doi: 10.1016/S0140-6736(16)30468-8. Epub 2016 May 18. PMID 27209146

DOCUMENTS (1):
  • Informed Consent Form (2022-05-22): https://cdn.clinicaltrials.gov/large-docs/47/NCT05568147/ICF_000.pdf